CLINICAL TRIAL: NCT00023309
Title: Combination of Lamivudine and Adefovir Dipivoxil for Treatment of Chronic Hepatitis B
Brief Title: Lamivudine and Adefovir to Treat Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marc Ghany, M.D., Principal Investigator, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010246; 01-DK-0246 (Other: NIHCC)
Record Dates: First submitted 2001-09-03; First posted 2001-09-03 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2014-07

CONDITIONS: HBV (Hepatitis B Virus); Hepatitis B; Hepatitis
Keywords: Adefovir Dipivoxil; Lamivudine; Nucleoside/Nucleotide Analogue; Chronic Hepatitis B; Hepatitis B Mutants; Liver Biopsy; Hepatitis B; Hepatitis; HBV; Liver
MeSH Terms: conditions — Hepatitis B; Hepatitis; Hepatitis B, Chronic | interventions — Lamivudine; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamivudine and adefovir (Experimental)
  Interventions: Drug: Lamivudine and adefovir
- Adefovir (Active Comparator)
  Interventions: Drug: Adefovir alone

INTERVENTIONS:
Drug: Lamivudine and adefovir — Lamivudine (100 mg/day) and adefovir (10 mg/day)
  Arms: Lamivudine and adefovir
Drug: Adefovir alone — Adefovir (10 mg/day)
  Arms: Adefovir

SUMMARY:
This study will evaluate the safety and effectiveness of lamivudine plus adefovir versus adefovir alone to treat chronic hepatitis B infection. The Food and Drug Administration has approved lamivudine for the treatment of hepatitis B. However, the drug is not effective in all patients, and many of those in whom it initially works develop resistance after 1 to 3 years. Adefovir is an experimental drug that inhibits replication of the hepatitis B virus (HBV). Adefovir used alone may be adequate to provide sustained suppression of the virus and improvement in liver disease. However combining two anti-viral agents may be superior to using one alone, similar to the strategy employed for the treatment of AIDS. This study will test whether the combination of lamivudine and adefovir is better than adefovir alone for the treatment of chronic hepatitis B.

Patients 18 years of age and older, who have been infected with HBV for at least 6 months, may be eligible for this study. Candidates may not have received lamivudine treatment in the past 6 months or prior treatment with adefovir and must not be taking other anti-viral treatments for their hepatitis. They will have a blood test to confirm HBV infection.

Participants will be admitted to the NIH Clinical Center for 2 to 3 days for a medical evaluation. One to 2 weeks after the evaluation, patients will be randomized to begin taking lamivudine and adefovir, or adefovir alone. Therapy will continue for at least 12 months. Follow-up clinic visits will be scheduled weekly for the first month, then every 4 to 8 weeks for the rest of the treatment period. Patients will be evaluated at the end of 1 year. Patients who have not improved with treatment will stop taking the treatment and will be evaluated in the clinic once every 4 weeks for another 6 months. Patients who show an improvement in their liver injury may continue taking lamivudine and adefovir or adefovir alone for 4 more years, as long as they continue to improve with the medication. Progress will be evaluated. If the test results show no continued improvement or are negative for hepatitis B antigens, therapy will be stopped.

Patients who continue treatment for 5 years will be readmitted at year 4 for another medical evaluation to assess the effects of treatment at that time. After the 5 years all patients will stop therapy at and be followed with regular clinic visits for at least 6 months.

DETAILED DESCRIPTION:
Aims: To assess the safety, antiviral activity and clinical benefit of the combination of lamivudine and adefovir dipivoxil vs adefovir alone in up to 80 patients with chronic hepatitis B for up to five years.

Background: Adefovir dipivoxil and lamivudine are oral antiviral agents that have been shown to have potent activity against HBV in vitro and in vivo. Both drugs have been used extensively in patients with HIV infection and more recently in controlled trials as monotherapy in patients with chronic hepatitis B. Lamivudine is currently approved as therapy of hepatitis B and has been evaluated extensively both as a one-year course of treatment as well as long-term continuous therapy. While lamivudine monotherapy induces a transient improvement in viral levels and liver histology, viral resistance develops in a large proportion of patients with re-appearance of HBV DNA in serum in high levels associated with mutations in the Tyrosine-methionine-aspartate-aspartate (YMDD) motif of the HBV polymerase gene and worsening of the hepatitis. Adefovir monotherapy, in contrast, has not been shown to be associated with development of viral resistance even when given for up to two years. When given as monotherapy for 1 year, adefovir leads to improvement in histology of hepatitis B in approximately 50% of patients. At present, the long-term efficacy of adefovir has not been shown.

Protocol: Up to 80 patients with chronic hepatitis B who have raised serum ALT (alanine aminotransferase) levels, HBV DNA in serum (above 1 million copies per ml by quantitative PCR) and active liver disease on liver biopsy will be enrolled and started on the combination of lamivudine (100 mg daily) and adefovir dipivoxil (10 mg daily) or adefovir alone (10 mg daily). Patients will be stratified into one of four groups of 20 patients for randomization: (A) Lamivudine naive and HBeAg positive, (B) Lamivudine naive and HBeAg negative (C) previous lamivudine therapy and HBeAg positive and (D) previous lamivudine therapy and HBeAg negative. Patients will be monitored carefully during therapy for adverse events, clinical symptoms and signs of liver disease, biochemical, and hematological parameters, and HBV serology at 2 to 4 week intervals. The primary endpoint of therapy will be a maintained combined response (a combination of virological, biochemical, and histological response) with major timing of end-points being at 1 and 4 years. Secondary endpoints will include loss of HBeAg, the individual types of maintained responses (virological, biochemical and histological), the development of lamivudine resistance, and improvement in symptom scores and quality of life assessments at 1 and 4 years.

Conclusions: This study will assess the effects of the combination of lamivudine and adefovir dipivoxil compared to adefovir alone in suppressing hepatitis B and prevention of lamivudine resistant mutants that arise during long-term therapy with lamivudine alone.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than 18 years and above, male or female

Known serum HBsAg positivity for at least 6 months

Detectable HBV-DNA in serum above 1 million copies per ml, as detected by quantitative PCR (Roche Cobas Assay)

Serum ALT (alanine aminotransferase) or AST (aspartate aminotransferase)levels above the upper limit of normal based on two determinations taken at least one month apart during the 6 months before entry

Liver biopsy within 2 years consistent with chronic hepatitis and with a histology activity index score (HAI) of 6 or more (out of a total possible score of 22) and an "Ishak" fibrosis score of at least 1 (out of a total possible score of 6). For patients with lamivudine resistance the liver biopsy may be performed either on or off lamivudine.

Written informed consent.

EXCLUSION CRITERIA:

Previous or current treatment with adefovir or tenofovir.

Co-infection with HDV (Hepatitis D Virus) as defined by the presence of both anti-HDV in serum and HDV antigen in liver

Co-infection with HCV (Hepatitis C Virus) as defined by the presence of both anti-HCV and HCV RNA in serum.

Co-infection with HIV (Human immunodeficiency virus) as defined by the presence of anti-HIV in serum.

Decompensated liver disease as defined by serum bilirubin greater than 2.5 mg%, prothrombin time of greater than 2 seconds prolonged, a serum albumin of less than 3.0 gm%, or a history of ascites, variceal bleeding, or hepatic encephalopathy.

Presence of other causes of liver disease (i.e., hemochromatosis, Wilson's disease, alcoholic liver disease, non-alcoholic steatohepatitis, alpha-1 antitrypsin deficiency)

A history of organ transplantation or in the absence of organ transplantation, any immunosuppressive therapy requiring the use of more than 5 mg of prednisone (or its equivalent) daily.

Significant systemic illnesses other than liver diseases including congestive heart failure, renal failure, chronic pancreatitis, diabetes mellitus with poor control that in the opinion of the investigators might interfere with therapy.

Pregnancy or inability to practice contraception in patients capable of bearing or fathering children

Pre-existing bone marrow suppression: White Blood Cells (WBC) less than 2,000 cells/mm(3), hematocrit less than 30%, or platelets less than 50,000 cells/mm(3).

History of clinically apparent pancreatitis or evidence of subclinical pancreatitis as shown by serum amylase values twice the upper limits of the normal range and abnormalities of the pancreas on CT or other imaging studies of the abdomen

Prior interferon treatment within 6 months of entry

Sensory or motor neuropathy apparent from medical history and physical examination

Creatinine clearance less than 50 ml/min or serum creatinine greater than 1.5 mg/dl; creatinine clearance will be determined on a 24 hour urine specimen. Accuracy of collection will be ensured by documenting appropriate total creatinine excretion in the 24 hour urine specimen (15 mg/kg) and correcting for the patient's age and gender.

Concurrent use of nephrotoxic agents (e.g., aminoglycosides, amphotericin B, vancomycin, foscarnet, cis-platinum, pentamidine, nonsteroidal anti-inflammatory agents) or competitors of renal tubular excretion (e.g., probenecid) within 2 months prior to study screening or the expectation that the subject will receive these during the course of the study

History of hypersensitivity to nucleoside/nucleotide analogues

Active ethanol/drug abuse/psychiatric problems that, in the investigator's opinion, might interfere with participation in the study

History of seizure disorder

History of renal tubular acidosis

History of malignancy or treatment for a malignancy within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-08; Primary Completion 2010-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghany Mark, MD, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Niederau C, Heintges T, Lange S, Goldmann G, Niederau CM, Mohr L, Haussinger D. Long-term follow-up of HBeAg-positive patients treated with interferon alfa for chronic hepatitis B. N Engl J Med. 1996 May 30;334(22):1422-7. doi: 10.1056/NEJM199605303342202. PMID 8618580
- [Background] Malik AH, Lee WM. Chronic hepatitis B virus infection: treatment strategies for the next millennium. Ann Intern Med. 2000 May 2;132(9):723-31. doi: 10.7326/0003-4819-132-9-200005020-00007. PMID 10787366
- [Background] Hoofnagle JH, di Bisceglie AM. The treatment of chronic viral hepatitis. N Engl J Med. 1997 Jan 30;336(5):347-56. doi: 10.1056/NEJM199701303360507. No abstract available. PMID 9011789
- [Derived] Ghany MG, Feld JJ, Zhao X, Heller T, Doo E, Rotman Y, Nagabhyru P, Koh C, Kleiner DE, Wright EC, Liang TJ, Hoofnagle JH. Randomised clinical trial: the benefit of combination therapy with adefovir and lamivudine for chronic hepatitis B. Aliment Pharmacol Ther. 2012 May;35(9):1027-35. doi: 10.1111/j.1365-2036.2012.05059.x. Epub 2012 Mar 26. PMID 22449251
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DK-0246.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-one patients were enrolled, twenty-two were randomized to receive the combination lamivudine and adefovir and nineteen to receive adefovir alone.
Groups:
- Lamivudine and Adefovir: Patients to receive combination lamivudine and adefovir, with lamivudine of 100 mg daily and adefovir of 10 mg daily
- Adefovir: Patients to receive adefovir alone (10 mg daily).
Period: Overall Study
Arm/Group | Lamivudine and Adefovir | Adefovir
Started | 22 | 19
Completed | 22 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lamivudine and Adefovir: Patients to receive combination lamivudine and adefovir
- Adefovir: Patients to receive adefovir alone
- Total: Total of all reporting groups
Arm/Group | Lamivudine and Adefovir | Adefovir | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14) | 45 (13) | 45 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 16 | 18 | 34
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9 | 8 | 17
  Asian | 9 | 10 | 19
  Black | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41
Treatment Naive [Number; unit: participants]
  Yes | 17 | 14 | 31
  No | 5 | 5 | 10
HBeAg positive [Number; unit: participants]
  Yes | 17 | 14 | 31
  No | 5 | 5 | 10
ALT [Mean (Standard Deviation); unit: IU/ml] — Alanine transaminase
  IU/ml | 183 (250) | 87 (56) | 139 (187)
HBV DNA Log 10 copies per ml [Mean (Standard Deviation); unit: log10(copies/ml)] — Hepatitis B virus DNA logarithm 10 copies per ml
  log10(copies/ml) | 8.1 (1.3) | 7.8 (1.6) | 8.0 (1.4)
HAI [Mean (Standard Deviation); unit: Units on a scale] — HAI Fibrosis score for liver histology, which has a range 0-18 and higher values represent a worse outcome
  Units on a scale | 8.1 (2.7) | 7.9 (2.4) | 8.0 (2.6)
Ishak [Mean (Standard Deviation); unit: Units on a scale] — Ishak Fibrosis Score, (range 0-6, where 0 = no fibrosis and 6 = cirrhosis)
  Units on a scale | 3.3 (1.7) | 2.4 (1.5) | 2.9 (1.6)
Cirrhosis [Number; unit: participants]
  Yes | 5 | 2 | 7
  No | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Maintained Combined Response (Virological, Biochemical and Histological Response).
Description: A maintained combined response was defined as a combination of a virological, biochemical and histological responses at weeks 48 and 192. A virological response was defined as a decrease in HBV DNA levels to undetectable by the Amplicor assay (<500 copies/mL). A biochemical response was defined as a decrease in serum ALT levels into the normal range (<41 U/L). A histological response was defined as a decrease in the HAI score by at least three points with no worsening of the Ishak fibrosis score.
Time Frame: 196 weeks from randomization
Population: The analysis was intention to treat. Patients with missing values at week 196 were treated as random missing. No imputation was applied.
Measure: Number; unit: participants
Arm/Group | Lamivudine and Adefovir | Adefovir
Number analyzed (Participants) | 22 | 19
participants
  Yes | 15 | 6
  No | 7 | 13
Statistical Analysis 1: Comparison: Lamivudine and Adefovir vs Adefovir; Null hypothesis: there is no difference in the treatment effect between the two groups; Test type: Superiority or Other; p = 0.0294, Fisher Exact

2. Secondary Outcome: HBeAg Loss at Week 196
Description: Loss of hepatitis B surface antigen (HBsAg) at week 196
Time Frame: Week 196 from randomization
Population: Analysis was intention to treat. Patients with missing values at timeframe of interest was taken as random missing. No imputation was applied.
Measure: Number; unit: participants
Arm/Group | Lamivudine and Adefovir | Adefovir
Number analyzed (Participants) | 17 | 14
participants
  Yes | 13 | 5
  No | 4 | 9
Statistical Analysis 1: Comparison: Lamivudine and Adefovir vs Adefovir; Null hypothesis: there is no difference in treatment effect at week 196; Test type: Superiority or Other; p = 0.0325, Fisher Exact

3. Secondary Outcome: Virological Response
Description: A virological response was defined as a decrease in HBV DNA levels to undetectable by the Amplicor assay (<500 copies/mL).
Time Frame: Week 196 from randomization
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Lamivudine and Adefovir | Adefovir
Number analyzed (Participants) | 22 | 19
participants
  Yes | 17 | 6
  No | 5 | 13
Statistical Analysis 1: Comparison: Lamivudine and Adefovir vs Adefovir; Null hypothesis: there is no difference in treatment effect at week 196; Test type: Superiority or Other; p = 0.0049, Fisher Exact

4. Secondary Outcome: Biological Response
Description: A biochemical response was defined as a decrease in serum ALT levels into the normal range (<41 U/L).
Time Frame: week 196 from randomization
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Lamivudine and Adefovir | Adefovir
Number analyzed (Participants) | 22 | 19
participants
  Yes | 21 | 12
  No | 1 | 7
Statistical Analysis 1: Comparison: Lamivudine and Adefovir vs Adefovir; Null hypothesis: there is no difference in treatment effect at week 196; Test type: Superiority or Other; p = 0.0157, Fisher Exact

5. Secondary Outcome: Histological Response
Description: A histological response was defined as a decrease in the HAI score by at least three points with no worsening of the Ishak fibrosis score.
Time Frame: week 196 from randomization
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Lamivudine and Adefovir | Adefovir
Number analyzed (Participants) | 18 | 10
participants
  Yes | 15 | 5
  No | 3 | 5
Statistical Analysis 1: Comparison: Lamivudine and Adefovir vs Adefovir; Null hypothesis: there is no difference in treatment effect at week 196; Test type: Superiority or Other; p = 0.0913, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Lamivudine and Adefovir | Adefovir
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No